CLINICAL TRIAL: NCT04119856
Title: Outgoing Lung Team - a Cross-sectorial and Preventive Intervention in Patients at Risk of Hospitalisation Due to Exacerbation of COPD
Brief Title: Outgoing Lung Team - a Cross-sectorial Intervention in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Outgoing Lung Team
Record Dates: First submitted 2019-10-07; First posted 2019-10-08 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-07

CONDITIONS: COPD; COPD Exacerbation
Keywords: Cross-sectorial; Hospitalization; Self-efficacy; Patient Involvement; Health Literacy; Anxiety
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Patient Participation; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Other): Affiliation with outgoing lung team
  * Instructions and teaching by the outgoing lung team.
  * Needs-based consultation at Dept. of Respiratory Diseases and Allergy.
  * Contact to the outgoing lung team in case of exacerbation of COPD.
  Interventions: Other: Affiliation with the outgoing lung team
- Control group (No Intervention): The usual practice
  * Scheduled consultations at Dept. of Respiratory Diseases and Allergy.
  * Contact to GP/doctor on call in case of exacerbation of COPD.

INTERVENTIONS:
Other: Affiliation with the outgoing lung team — The work of the outgoing lung team takes place in the patient's home and involves the following:
  * The outgoing lung team teaches the patients, relatives and primary care staff about symptoms, treatments and instructions related to COPD.
  * The patients, relatives and primary care staff can contact the outgoing lung team by telephone day and night.
  * The patients report symptoms and measurements to the outgoing lung team using telemedicine as patient reported outcomes.
  * The outgoing lung team initiates appropriate treatment by telephone or a home visit. The outgoing lung team always consults a doctor from the Department of Respiratory Diseases and Allergy before initiating treatment.
  * The outgoing lung team initiates acute consultations at Department of Respiratory Diseases and Allergy based on patient reported outcomes, home visit or telephone call.
  Arms: Intervention group

SUMMARY:
This study examines the effects of the work of an outgoing lung team in the Municipality of Aarhus, Denmark to patients with COPD (Chronic obstructive pulmonary disease) at risk of exacerbation of COPD.

The outgoing lung team is a cross-sectorial team of nurses and doctors from Department of Respiratory Diseases and Allergy at Aarhus University Hospital and nurses from the Acute Team in the Municipality of Aarhus.

The work of the outgoing lung team takes place in the patient's home and involves the following:

* The outgoing lung team teaches the patients, relatives and primary care staff about symptoms, treatments and instructions related to COPD.
* The patients, relatives and primary care staff can contact the outgoing lung team by telephone day and night.
* The outgoing lung team initiates appropriate treatment by telephone or a home visit in consultation with a doctor.
* The patients report symptoms and measurements to the outgoing lung team using telemedicine solutions (AmbuFlex).
* The outgoing lung team initiates acute consultations at Department of Respiratory Diseases and Allergy based on patient reported outcomes, home visit or telephone call.

Half of the participants are affiliated to the outgoing lung team, while the other half are not, and continue their usual practice by contacting the general practitioners in case of exacerbation of COPD.

The main hypothesis of the project is that outgoing lung team has a positive impact on continuity of care across sectors in the Danish healthcare system for patients with COPD. More specifically the hypotheses are:

1. Affiliation to the outgoing lung team reduces admissions, readmissions, length of hospital stay and outpatient consultations.
2. Affiliation to the outgoing lung team reduces anxiety and depression and increases patient involvement, and improves patients' health status and self-efficacy.
3. Affiliation to the outgoing lung team increases patients' level of health literacy.

DETAILED DESCRIPTION:
Background

Worldwide, COPD is a major cause of morbidity and mortality and is currently the fourth leading cause of death and projected to be the third leading cause of death by 2020. In 2010, the estimated number of COPD cases worldwide was 384 million with a prevalence of 11% (95% confidence interval: 8,4%-15,0%).

COPD is characterised by airway obstruction due to inflammation and destruction of lung tissue. The disease causes breathlessness, cough, mucus and frequent respiratory infections and leads to decreased lung function. COPD often affects patients' quality of life negatively as many experience anxiety because of breathlessness. Breathing difficulties reduce patients' level of activity and can lead to social isolation. In Denmark, it is estimated that 320,000 Danes have COPD. In 2018, the number of admissions due to COPD in Denmark was 34,961 with a readmission rate (new hospitalisation within 30 days after the last hospitalisation) of 19% and a 30-day mortality rate of 11%.There were 49,424 outpatient visits due to COPD in Denmark in 2018, and approximately 5,500 annual deaths where COPD is the direct or contributory cause.

It is estimated that the total annual treatment costs for patients with COPD in Denmark amount to approximately DKK 3,345 billion, and most of these costs are related to acute admissions.

Previous research shows that patients with COPD experience not being offered the same quality of treatment as other chronic patients. Furthermore, patients with COPD report that they are not taken seriously by healthcare professionals, which induces insecurity.

As patients with COPD constitute a large group in both the primary and secondary care, we intend to improve the collaboration between the two sectors based on patients´ preferences. The patients emphasized the importance of having the possibility to contact a specialised respiratory nurse 24-7. Patients reported that they preferred education to take place close to home, as transportation to hospital or the community support centre for older people were both mentally and physically straining.

Research showed that home visits by a respiratory nurse from the hospital reduce admissions and readmissions. Furthermore, research showed that home visits by the nurses in primary care also decrease admissions and readmissions. Some of the interventions were treatment at home and some comprised education regarding management of acute exacerbations and observations of symptoms, inhalation, smoking cessation, nutrition etc.

The interventions consisted of collaboration between primary care nurses and the general practitioners (GPs), and in other interventions primary care nurses were supervised by the specialist respiratory nurses at the hospital often by phone or at joint visits in the patients' home.

Home visits after discharge paid by a respiratory nurse and interdisciplinary cooperation showed that patients with COPD felt safe and comforted and were motivated to make changes to achieve better health.

However, other studies showed that education improved patients' knowledge but it did not prevent readmissions.

So far, no studies have been performed investigating cross-sectorial collaboration with a lung team and preventive intervention in patients at risk of hospitalisation due to exacerbation of COPD.

Department of Respiratory Diseases and Allergy at Aarhus University Hospital, Denmark and the Acute Team in the Municipality of Aarhus, Denmark started a pilot project from September 2015 until October 2016. The project concerned establishment of an outgoing lung team comprised by a team of nurses from both the primary and secondary sector. The aim was to increase knowledge and competences among patients, relatives and staff in relation to care and treatment, to reduce the rate of hospitalisation and readmission and to evaluate the impact of the outgoing lung team on participants' health status. The pilot project had several limitations 1) It was only possible to evaluate the effect of the outgoing lung team during six months. We were thus unable to evaluate variety over the year which may have impacted on the number of hospitalisations, readmissions and episodes of exacerbation. 2) The pilot project had no control group. We thus wanted to qualify the project by using a randomised controlled trial design.

We also wanted to examine the impact of the outgoing lung team on the level of patient involvement, anxiety, depression and health literacy. Health literacy is linked to literacy and entails people's knowledge, motivation and competences to access, understand, appraise and apply health information in order to make judgements and take decisions in everyday life concerning health care, disease prevention and health promotion to maintain or improve quality of life during the life course. Studies show that patients with COPD have lower levels of health literacy compared with people with no chronic diseases. Increasing the level of health literacy in this population would thus be relevant.

Furthermore, we wished to examine the effect of the outgoing lung team on patients' health status, their experiences of being affiliated to the outgoing lung team as well as their self-efficacy.

Objective

The aim is to examine the effects of the work of an outgoing lung team in the Municipality of Aarhus to patients with COPD at risk of exacerbation of COPD.

Hypothesis

The main hypothesis is that outgoing lung team has a positive impact on continuity of care across sectors in the Danish healthcare system for patients with COPD. To examine this we have three subhypotheses.

1. Affiliation to the outgoing lung team reduces admissions, readmissions, length of hospital stay and outpatient consultations.
2. Affiliation to the outgoing lung team reduces anxiety and depression and increases patient involvement, and improves patients' health status and self-efficacy.
3. Affiliation to the outgoing lung team increases patients' level of health literacy.

Materials and method

Setting and location

The outgoing lung team is a cross-sectorial team of nurses and doctors from Department of Respiratory Diseases and Allergy at Aarhus University Hospital in Denmark and nurses from the Acute Team in the Municipality of Aarhus in Denmark. The outgoing lung team intends to preserve, detect, diagnose and treat patients with an exacerbation of COPD. The outgoing lung team is physically located at the office of the Acute Team; in this office knowledge sharing and upgrading of skills take place.

The work of the outgoing lung team takes place in the patient's home and involves the following:

* The outgoing lung team teaches the patients, relatives and primary care staff about symptoms, treatments and instructions related to COPD.
* The patients, relatives and primary care staff can contact the outgoing lung team by telephone day and night.
* The patients report symptoms and measurements to the outgoing lung team using telemedicine solutions, also known as patient reported outcomes.
* The outgoing lung team initiates appropriate treatment by telephone or a home visit. The outgoing lung team always consults a doctor from the Department of Respiratory Diseases and Allergy before initiating treatment.
* The outgoing lung team initiates acute consultations at Department of Respiratory Diseases and Allergy based on patient reported outcomes, home visit or telephone call.

Doctors at Department of Respiratory Diseases and Allergy are responsible for the medical treatment as long as the patient participates in the project. The GPs in the Municipality of Aarhus have agreed to this. The GPs can refer patients to the project and some of them participate in a project advisory board.

Study design

The project is designed as a mixed-method study based on a randomised controlled trial with an intervention group connected to the outgoing lung team and a control group attending the standard pathway programme at Department of Respiratory Diseases and Allergy at Aarhus University Hospital, Denmark.

Sample size

Based on a retrospective sample of admissions related to COPD in the period from February to August 2014-2016, an expected decrease in length of hospital stay can be calculated as the outgoing lung team was introduced in 2016. Mean number of admission days in the retrospective sample followed a normal distribution after logarithmic transformation, as assessed by histograms. Number of admission days (geometric mean) was 5.69 (95% CI: 2.78-11.6) in 2014-2015, and 4.50 (2.62-7.76) in 2016. Based on these numbers, the power calculation resulted in inclusion of 64 patients in the intervention and control group, respectively to be able to demonstrate a significant difference with a power of 80% and at a significance level of 5%.

In the pilot project the withdrawal was 23%. With an estimated withdrawal at 23% we will need 83 patients in each group.

Missing data

After one year, we contact all participants and arrange a plan for answering the questionnaires. The missing data, will be registered in Stata and mentioned in the study.

Analysis

Data will be statistically analysed both descriptive and analytically. Correlations and significant factors as lung function, gender, age etc. will be examined and significant differences between the two groups (intervention group and control group) in the studies which may have an impact on results.

To identify predictors of the impact on the dependent variable we will use bivariate x 2 test and calculation of odds ratios, multiple logistic regression and logarithmic data. The statistical analysis will be performed in Stata 16.

Qualitative data from the interviews in will be transcribed and analysed based on meaning condensation analysis.

Ethics

Ethical approval will be obtained from Central Denmark Region Committees on Health Research Ethics and approval of data archives and storage will be obtained from the Danish Data Protection Agency in Central Denmark Region in RedCap. All collected personal data will be anonymised, processed, analysed and stored in accordance with the Danish Data Protection Agency. All participants will receive oral and written information. Patients who agree to participate will provide written informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Citizens of the Municipality of Aarhus
2. FEV1 <50% predicted and at least one hospitalisation due to COPD and/or two tablet-treated episodes of exacerbation (prednisolone and /or antibiotics) within the last year
3. Special needs due to anxiety, dyspnea etc. that cause frequent hospitalisations

Exclusion Criteria:

1. Participation in the pilot project
2. Inability to speak, read and understand Danish
3. Severe cognitive disability and thus inability to understand and fill in questionnaires (e.g. dementia)
4. No wish to participate in the project

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Change in admissions and re-admissions. | One year. From date of randomization and after one year.
  Data from the patients records.
Length of hospitalisation related to COPD. | One year. From date of randomization and after one year
  Data from the patients records.

SECONDARY OUTCOMES:
Number of outpatient consultations related COPD. | One year. From date of randomization and after one year.
  Data from the patients records.
Measure level of patient involvement | One year. From date of randomization and after one year.
  Self reported level of patient involvement. The questionnaire PACIC (Patient Assessment of Chronic Illness Care) comprised of 20-items. Each item is scored "Never", "Usually not", "Sometimes" "Usually" or "Always"
Change in health status | One year. From date of randomization and after one year.
  Self reported health status. The questionnaire CAT (COPD Assessment Test) comprised of 8 items. Each item is scored 0-5 (O = never, and 5 = always)
Change in quality of life | One year. From date of randomization and after one year.
  Self reported data based on the questionaire EQ-5D-3L (Euro-quality of life group- 5 dimensions- 3 level). Each item is scores 1-3 (1= No problems, 3= Many problems)
Change in anxiety and depression | One year. From date of randomization and after one year.
  Self reported data based on the questionaire HADS (Hospital Anxiety and Depression Scale). It consists of 14 items. Each items is scored 1-4 (1 = Most of the time/ definitely to 4= very rare/ definitely not)
Change in level of health literacy | One year. From date of randomization and after one year.
  Self reported data based on the questionaire HLQ (Health Literacy Questionnaire). It comprises of 9 domains. In this study we use 3 domains and it consists of 15 items. 1 domain comprised of 5 items, and each item is scored from "totally not agree" to " not agree", "agree" and "totally agree". The two other domains comprises in total of 10 domains, where each item is scored from "Always difficult", "Often difficult", "Sometimes difficult", "Often easy" and "Always easy".
Change in self-efficacy | One year. From date of randomization and after one year.
  Self reported data based on the questionaire CSES (COPD Self-Efficacy Scale). It comprises of 34 items, and each item is scores from "very sure", "pretty Sure", "partly sure", "not very sure" and definitely not sure"
Experiences of affiliation with the outgoing lung team. | One time after, they have been affiliated with the outgoing lung team for at least 7 month.
  Interviews with patients who have been affiliated with the outgoing lung team.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit R Iversen, Ph.d.-stud., Study Director — Department of Respiratory Diseases and Allergy, Aarhus University Hospital
Locations (1):
- Department of Respiratory Diseases and Allergy, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Global Initiative for Chronic Obstructive Lung Disease. Global Strategy for Diagnosis, Management, and Prevention of COPD - 2019. 2019; Available at: https://goldcopd.org/wp-content/uploads/2018/11/GOLD-2019-v1.7-FINAL-14Nov2018-WMS.pdf. Accessed 15.04, 2019.
- [Background] Sundhedsstyrelsen. Anbefalinger for tværsektorielle forløb for mennesker med KOL. 2017; Available at: https://www.sst.dk/da/udgivelser/2017/~/media/8365DCEC9BB240A0BD6387A81CBDBB49.ashx. Accessed 04.07, 2017.
- [Background] Dansk Register for Kronisk Obstruktiv Lungesygdom. Appendiks til National årsrapport 2018. 2019; Available at: https://www.sundhed.dk/content/cms/90/4690_appendix_drkol-aarsrapport-2018_05052019_offentlig.pdf. Accessed 12.08, 2019.
- [Background] Dansk Register for Kronisk Obstruktiv Lungesygdom. National årsrapport 2018. 2019; Available at: https://www.sundhed.dk/content/cms/90/4690_drkol-aarsrapport-2018_offentlig.pdf. Accessed 12.08, 2019.
- [Background] Witzel S, Nielsen PB, Jensen M. Patienternes perspektiv på kronisk sygdom - Oplevelser på tværs af sundhedsvæsenet i Region Midtjylland. CFK - Folkesundhed og Kvalitetsudvikling. 2012; Available at: http://www.defactum.dk/publikationer/ShowPublication?id=421&pageId=309986. Accessed 05.07, 2016.
- [Background] Martin HM, Borst L. Sammenhæng i tværsektorielle KOL - forløb. En undersøgelse af patient er og pårørendes oplevelser. KORA - Det Nationale Institut for Kommuners og Regioners Analyse og Forskning. 2013; Available at: https://www.vive.dk/media/pure/9106/2043881. Accessed 05.07, 2019.
- [Background] Rasmussen L, Ølsgaard G. Forslag til kvalitetsforbedringer fra patienter og fagpersoner i indsatsen for kronisk syge - en opfølgning på rapporten "Patientens perspektiv på kronisk sygdom". CFK - Folkesundhed og Kvalitetsudvikling. 2014; Available at: http://www.defactum.dk/publikationer/ShowPublication?id=435&pageId=309986. Accessed 05.07, 2016.
- [Background] Haggerty MC, Stockdale-Woolley R, Nair S. Respi-Care. An innovative home care program for the patient with chronic obstructive pulmonary disease. Chest. 1991 Sep;100(3):607-12. doi: 10.1378/chest.100.3.607. PMID 1889241
- [Background] Pearson S, Inglis SC, McLennan SN, Brennan L, Russell M, Wilkinson D, Thompson DR, Stewart S. Prolonged effects of a home-based intervention in patients with chronic illness. Arch Intern Med. 2006 Mar 27;166(6):645-50. doi: 10.1001/archinte.166.6.645. PMID 16567604
- [Background] Transition reduced readmission rate for COPD patients. Hosp Case Manag. 2010 May;18(5):71-3. No abstract available. PMID 20449991
- [Background] Ward S, Barnes H, Ward R. Evaluating a respiratory intermediate care team. Nurs Stand. 2005 Oct 12-18;20(5):46-50. doi: 10.7748/ns2005.10.20.5.46.c3975. PMID 16255486
- [Background] Rea H, McAuley S, Stewart A, Lamont C, Roseman P, Didsbury P. A chronic disease management programme can reduce days in hospital for patients with chronic obstructive pulmonary disease. Intern Med J. 2004 Nov;34(11):608-14. doi: 10.1111/j.1445-5994.2004.00672.x. PMID 15546454
- [Background] Matsumura T, Takarada K, Oki Y, Fujimoto Y, Kaneko H, Ohira M, Ishikawa A. Long-term Effect of Home Nursing Intervention on Cost and Healthcare Utilization for Patients with Chronic Obstructive Pulmonary Disease: A Retrospective Observational Study. Rehabil Nurs. 2015 Nov-Dec;40(6):384-9. doi: 10.1002/rnj.189. Epub 2014 Nov 25. PMID 25425110
- [Background] Spiliopoulos N, Donoghue J, Clark E, Dunford M. Outcomes from a Respiratory Coordinated Care Program (RCCP) providing community-based interventions for COPD patients from 1998 to 2006. Contemp Nurse. 2008 Dec;31(1):2-8. doi: 10.5172/conu.673.31.1.2. PMID 19117496
- [Background] Cox K, Macleod SC, Sim CJ, Jones AW, Trueman J. Avoiding hospital admission in COPD: impact of a specialist nursing team. Br J Nurs. 2017 Feb 9;26(3):152-158. doi: 10.12968/bjon.2017.26.3.152. PMID 28185492
- [Background] Titova E, Steinshamn S, Indredavik B, Henriksen AH. Long term effects of an integrated care intervention on hospital utilization in patients with severe COPD: a single centre controlled study. Respir Res. 2015 Feb 3;16(1):8. doi: 10.1186/s12931-015-0170-1. PMID 25645122
- [Background] Lee G, Pickstone N, Facultad J, Titchener K. The future of community nursing: Hospital in the Home. Br J Community Nurs. 2017 Apr 2;22(4):174-180. doi: 10.12968/bjcn.2017.22.4.174. PMID 28414540
- [Background] Davison AG, Monaghan M, Brown D, Eraut CD, O'Brien A, Paul K, Townsend J, Elston C, Ward L, Steeples S, Cubitt L. Hospital at home for chronic obstructive pulmonary disease: an integrated hospital and community based generic intermediate care service for prevention and early discharge. Chron Respir Dis. 2006;3(4):181-5. doi: 10.1177/1479972306070074. PMID 17190120
- [Background] Hermiz O, Comino E, Marks G, Daffurn K, Wilson S, Harris M. Randomised controlled trial of home based care of patients with chronic obstructive pulmonary disease. BMJ. 2002 Oct 26;325(7370):938. doi: 10.1136/bmj.325.7370.938. PMID 12399344
- [Background] Zwar NA, Hermiz O, Comino E, Middleton S, Vagholkar S, Xuan W, Wilson SF, Marks GB. Care of patients with a diagnosis of chronic obstructive pulmonary disease: a cluster randomised controlled trial. Med J Aust. 2012 Oct 1;197(7):394-8. doi: 10.5694/mja12.10813. PMID 23025736
- [Background] Leine M, Wahl AK, Borge CR, Hustavenes M, Bondevik H. Feeling safe and motivated to achieve better health: Experiences with a partnership-based nursing practice programme for in-home patients with chronic obstructive pulmonary disease. J Clin Nurs. 2017 Sep;26(17-18):2755-2764. doi: 10.1111/jocn.13794. Epub 2017 May 17. PMID 28252816
- [Background] World Health Organization Europe. Health Literacy - The solid facts. 2013; Available at: http://www.euro.who.int/__data/assets/pdf_file/0008/190655/e96854.pdf?ua=1. Accessed 01.03, 2017.
- [Background] Friis K, Jensen ML, Lasgaard M, Maindal HT. Sundhedskompetence blandt personer med kronisk sygdom. Region Midtjylland CFK - Folkesundhed og Kvalitetsudvikling. 2015; Available at: https://www.rm.dk/siteassets/om-os/aktuelt/nyheder/sundhedskompetence_kronisk_sygdom_2015_temaanalyse.pdf. Accessed 13.07, 2016.
- [Background] Kvale S, Brinkmann S. Interview : det kvalitative forskningsinterview som håndværk. 3rd ed. København: Hans Reitzel; 2015.
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686